CLINICAL TRIAL: NCT03818711
Title: Communication and Coping: Addressing Mothers' Needs to Improve Outcomes in Adolescents With T1D
Brief Title: Communication and Coping for Mothers of Adolescents With Type 1 Diabetes
Acronym: T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Sarah Jaser, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 171940
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication & Coping Intervention (Experimental): A cognitive behavioral intervention for mothers of adolescents with type 1 diabetes to improve coping and the quality of parental involvement.
  Interventions: Behavioral: Communication & Coping Intervention
- Education & Check Ins (Active Comparator): The comparison group receives educational materials on diabetes management and phone calls, as well as access to a secret Facebook group with daily posts on diabetes management.
  Interventions: Behavioral: Education & Check Ins

INTERVENTIONS:
Behavioral: Communication & Coping Intervention — Mothers receive a treatment manual and participate in individual phone calls aimed at reducing depressive symptoms and improving the quality of parental involvement. A concurrent secret Facebook group will have daily posts to reinforce concepts.
  Arms: Communication & Coping Intervention
Behavioral: Education & Check Ins — Mothers receive educational materials and participate in individual phone calls related to these materials. A concurrent secret Facebook group will have daily educational posts.
  Arms: Education & Check Ins

SUMMARY:
Mothers of adolescents with type 1 diabetes experience high levels of depressive symptoms, which impair their ability to monitor and manage diabetes treatment effectively. Further, maternal depressive symptoms are one of the strongest predictors of negative outcomes in adolescents, including deteriorating glycemic control, problems with adherence, poorer quality of life, and greater risk for depression. Given that adolescents are a high-risk population for suboptimal glycemic control - with only 17% meeting treatment goals - there is a critical need for novel interventions to improve outcomes in adolescents with T1D. Yet, previous behavioral interventions for youth with diabetes have had only modest effects on glycemic control, and none have directly targeted maternal depressive symptoms.

Building on effective interventions to treat depression in adults, and our own pilot work in this population, the proposed study will use a rigorous approach to evaluate the efficacy of a cognitive-behavioral intervention for mothers of adolescents with type 1 diabetes to promote the use of adaptive coping strategies and positive parenting practices. The aims of this study are to: 1) evaluate the effects of the Communication & Coping intervention on diabetes-related outcomes; 2) evaluate the effects of the Communication & Coping intervention on psychosocial outcomes; and 3) explore the differential impact of the intervention across demographic factors. Mothers who are randomized to the Communication & Coping Intervention will receive individual cognitive-behavioral therapy sessions by phone, as well as access to a Facebook group to augment the material covered in calls and provide social support. Mothers randomized to the Attention Control condition will receive educational materials and phone check-ins, as well as a Facebook group with educational posts. Adolescents and their mothers will be assessed at baseline and again post-intervention, at 3 months, 6 months, and 12 months.

DETAILED DESCRIPTION:
Mothers of adolescents with type 1 diabetes experience high levels of depressive symptoms, which impair their ability to monitor and manage diabetes treatment effectively. The regimen recommended for type 1 diabetes is complex and demanding, and caregivers - especially mothers - experience stress related to the burden of treatment management. This stress is associated with increased risk for psychosocial problems in caregivers, with rates of clinically significant depressive symptoms evident in up to 61% of parents. Further, maternal depressive symptoms are one of the strongest predictors of negative outcomes in adolescents, including deteriorating glycemic control, problems with adherence, poorer quality of life, and greater risk for depression. Given that adolescents are a high-risk population for suboptimal glycemic control - with only 17% meeting treatment goals - there is a critical need for novel interventions to improve outcomes in adolescents with T1D. Yet, previous behavioral interventions for youth with diabetes have had only modest effects on glycemic control, and none have directly targeted maternal depressive symptoms. Responding to the American Diabetes Association's call to address the psychosocial needs of people with diabetes and their family members, the proposed project has the potential to improve outcomes in both adolescents with type 1 diabetes and their mothers.

Building on effective interventions to treat depression in adults, and our own pilot work in this population, the proposed study will use a rigorous approach to evaluate the efficacy of a cognitive-behavioral intervention for mothers of adolescents with type 1 diabetes to promote the use of adaptive coping strategies and positive parenting practices. The aims of this study are to: 1) evaluate the effects of the Communication & Coping intervention on diabetes-related outcomes; 2) evaluate the effects of the Communication & Coping intervention on psychosocial outcomes; and 3) explore the differential impact of the intervention across demographic factors. Mothers who are randomized to the Communication & Coping Intervention will receive individual cognitive-behavioral therapy sessions by phone, as well as access to a Facebook group to augment the material covered in calls and provide social support. Mothers randomized to the Attention Control condition will receive educational materials and phone check-ins, as well as a Facebook group with educational posts. Adolescents and their mothers will be assessed at baseline and again post-intervention, at 3 months, 6 months, and 12 months. We hypothesize that the adolescents of mothers who receive the intervention will demonstrate improvements in diabetes outcomes (i.e., glycemic control, adherence), as well as psychosocial outcomes (i.e., improved quality of life, fewer depressive symptoms) compared to those in the attention control condition. This approach is innovative by targeting maternal depressive symptoms and the quality of parental involvement in mothers of adolescents with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Female caregiver of an adolescent with type 1 diabetes
* Adolescent age 11-17
* Adolescent diagnosed with type 1 diabetes for at least 12 months
* Caregiver reports mild to moderate depressive symptoms (PHQ-9 score of 5-19) OR OR caregiver reports diabetes distress (Parent/Teen Relationship Distress Subscale score of 2 or higher)
* English speaking

Exclusion Criteria:

* Caregiver reports minimal depressive symptoms (PHQ-9 score less than 5)
* Caregiver reports severe depressive symptoms (PHQ-9 score 20 or higher)
* Caregiver reports history of severe psychopathology (bipolar disorder or schizophrenia)
* Caregiver reports that adolescent has history of severe psychopathology (bipolar disorder or schizophrenia)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female caregiver
Enrollment: 302 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Jaser, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from the Children's Diabetes Program at Vanderbilt, as well as the Vanderbilt Research Notifications Distribution List.
Pre-assignment Details: Caregiver-adolescent dyads were enrolled and randomized. After enrollment, maternal caregiver participants were required to connect to the study Facebook account prior to randomization.
  Protocol Enrollment, Number Started, and Completed reflect participants. 3 dyads were enrolled but not randomized: Two caregivers completed baseline data but did not connect to the study Facebook account.
  One dyad consented and started baseline surveys but decided not to continue.
Period: Baseline Through Intervention
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Started | 150 | 152
Caregivers | 75 | 76
Adolescents | 75 | 76
Completed | 148 | 150
Not Completed | 2 | 2
Period: 3-month Data Collection
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Started | 148 | 150
Caregiver | 74 | 75
Adolescent | 74 | 75
Completed | 144 | 148
Not Completed | 4 | 2
Period: 6-month Data Collection
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Started | 144 | 148
Caregiver | 72 | 74
Adolescent | 72 | 74
Completed | 144 | 142
Not Completed | 0 | 6
Period: 12-month Data Collection
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Started | 144 | 142
Caregiver | 62 | 64
Adolescent | 59 | 62
Completed | 121 | 126
Not Completed | 23 | 16

BASELINE CHARACTERISTICS:
Population: Participants were maternal caregiver-adolescent dyads
Groups:
- Total: Total of all reporting groups
Arm/Group | Communication & Coping Intervention | Education & Check Ins | Total
Number analyzed (Participants) | 150 | 152 | 302
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Caregiver age analyzed separately from adolescent age.
  years
    Caregiver Age: number analyzed (Participants) | 75 | 76 | 151
    Caregiver Age | 42 [39 to 47] | 41 [38 to 47] | 42 [38 to 47]
    Adolescent Age: number analyzed (Participants) | 75 | 76 | 151
    Adolescent Age | 14 [13 to 16] | 14 [12 to 16] | 14 [12 to 16]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were caregiver-adolescent dyads.
  Participants
    Caregiver Sex: number analyzed (Participants) | 75 | 76 | 151
    Caregiver Sex: Female | 75 | 76 | 151
    Caregiver Sex: Male | 0 | 0 | 0
    Adolescent Sex: number analyzed (Participants) | 75 | 76 | 151
    Adolescent Sex: Female | 45 | 39 | 84
    Adolescent Sex: Male | 30 | 37 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of caregivers and adolescents were analyzed separately. Population: Ethnicity of caregivers and adolescents were analyzed separately.
  Participants
    Maternal Caregiver Ethnicity: number analyzed (Participants) | 75 | 76 | 151
    Maternal Caregiver Ethnicity: Hispanic or Latino | 2 | 2 | 4
    Maternal Caregiver Ethnicity: Not Hispanic or Latino | 73 | 74 | 147
    Maternal Caregiver Ethnicity: Unknown or Not Reported | 0 | 0 | 0
    Adolescent Ethnicity: number analyzed (Participants) | 75 | 76 | 151
    Adolescent Ethnicity: Hispanic or Latino | 3 | 2 | 5
    Adolescent Ethnicity: Not Hispanic or Latino | 72 | 74 | 146
    Adolescent Ethnicity: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of caregivers and adolescents were analyzed separately. Population: Race of caregivers and adolescents analyzed separately.
  Participants
    Maternal Caregiver Race: number analyzed (Participants) | 75 | 76 | 151
    Maternal Caregiver Race: American Indian or Alaska Native | 0 | 0 | 0
    Maternal Caregiver Race: Asian | 0 | 0 | 0
    Maternal Caregiver Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Maternal Caregiver Race: Black or African American | 5 | 7 | 12
    Maternal Caregiver Race: White | 68 | 69 | 137
    Maternal Caregiver Race: More than one race | 2 | 0 | 2
    Maternal Caregiver Race: Unknown or Not Reported | 0 | 0 | 0
    Adolescent Race: number analyzed (Participants) | 75 | 76 | 151
    Adolescent Race: American Indian or Alaska Native | 0 | 0 | 0
    Adolescent Race: Asian | 0 | 0 | 0
    Adolescent Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescent Race: Black or African American | 5 | 9 | 14
    Adolescent Race: White | 63 | 65 | 128
    Adolescent Race: More than one race | 6 | 2 | 8
    Adolescent Race: Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — Population: Region of Enrollment for Caregivers only
  participants
    United States: number analyzed (Participants) | 75 | 76 | 151
    United States | 75 | 76 | 151
Region of Enrollment [Number; unit: participants] — Region of Enrollment for Adolescents Only
  participants
    United States | 75 | 76 | 151
Marital Status [Count of Participants; unit: Participants] — Marital status only analyzed for caregiver participants (not adolescents). Population: Marital status only analyzed for caregiver participants (not adolescents).
  Participants
    number analyzed (Participants) | 75 | 76 | 151
    Married/Partnered | 60 | 62 | 122
    Single/Divorced/Widowed | 15 | 14 | 29
Household Income [Count of Participants; unit: Participants] — Household income was only analyzed for caregiver participants (not adolescents) Population: Two caregivers did not provide information on income.
  Participants
    <$19,999: number analyzed (Participants) | 75 | 76 | 151
    <$19,999 | 4 | 4 | 8
    $20-$39,999: number analyzed (Participants) | 75 | 76 | 151
    $20-$39,999 | 5 | 8 | 13
    $40-$59,999: number analyzed (Participants) | 75 | 76 | 151
    $40-$59,999 | 13 | 11 | 24
    $60-$79,999: number analyzed (Participants) | 75 | 76 | 151
    $60-$79,999 | 14 | 13 | 27
    $80-$99,999: number analyzed (Participants) | 75 | 76 | 151
    $80-$99,999 | 11 | 12 | 23
    $100,000 or more: number analyzed (Participants) | 75 | 76 | 151
    $100,000 or more | 27 | 27 | 54
    Missing: number analyzed (Participants) | 75 | 76 | 151
    Missing | 1 | 1 | 2
Hemoglobin A1c [Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin] — Hemoglobin A1c measures the amount of glucose attached to hemoglobin. It is assessed as part of regular diabetes clinic visits. The target is <7.0%. Population: A1c only collected from adolescents participants (not caregivers), since adolescents had type 1 diabetes.
  percentage of glycated hemoglobin
    number analyzed (Participants) | 75 | 76 | 151
    (all) | 8.2 [7.2 to 10.4] | 8.7 [7.8 to 10.1] | 8.5 [7.4 to 10.2]

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control (A1C)
Description: Hemoglobin A1c measured as part of clinic visit indicates the amount of glucose attached to hemoglobin.
Time Frame: 12 months
Population: Only adolescents participants have the A1C value.
Measure: Median (Inter-Quartile Range); unit: Percentage of glycated hemoglobin
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 70 | 71
Percentage of glycated hemoglobin | 8.4 [7.3 to 10.2] | 8.5 [7.4 to 9.8]

2. Secondary Outcome: Maternal Depressive Symptoms
Description: Depressive symptoms measured using the Patient Health Questionnaire (PHQ-9), a 9-item measure. Scores range from 0-27; scores 0-4 indicate minimal depression, scores 5-9 indicate mild depression, scores 10-14 indicate moderate depression, scores 15-19 indicate moderately severe depression, and scores 20-27 indicate severe depression.
Time Frame: 3 months
Population: Only maternal caregiver participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 69
score on a scale | 6.4 (4.6) | 5.1 (4.6)

3. Secondary Outcome: Mothers' Diabetes Distress
Description: Parent Diabetes Distress Scale (PDDS) is a measure consisting of 20 items to rate diabetes-related stress for parents of children with type 1 diabetes. A mean total score will be calculated, ranging from 0-5, with higher scores indicating greater distress.
Time Frame: 3 months
Population: Only maternal caregiver participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 69
score on a scale | 1.58 (.80) | 1.72 (.84)

4. Secondary Outcome: Adolescent Psychosocial Functioning - Parent Report
Description: Child Behavior Checklist (CBCL) is a parent-reported measure of behavior problems in children ages 6-18. Raw scores are converted to age- and sex-normed T-Scores (mean = 50, SD = 10). Higher scores indicate greater problem behaviors.
Time Frame: 3 months
Population: Only maternal caregiver participants completed this measure.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 47 | 49
T-Score
  Internalizing Problems | 55.4 (8.7) | 57.3 (12.6)
  Externalizing Problems | 51.2 (9.9) | 52.4 (10.2)
  Depressive Problems | 58.5 (7.9) | 60.8 (10.1)

5. Secondary Outcome: Adolescent Psychosocial Functioning - Self Report
Description: Youth Self Report (YSR) is a measure of self-reported behavior problems in youth ages 11-18. The Child Behavior Checklist was completed by caregivers as a proxy report of adolescent's behaviors. Raw scores are converted to age- and sex-normed T-Scores (mean = 50, SD = 10). Higher scores indicate greater problem behaviors.
Time Frame: 3 months
Population: Only adolescent participants completed this measure.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 43 | 45
T-Score
  Internalizing Problems | 53.6 (12.3) | 54.4 (12.5)
  Externalizing Problems | 48.9 (10.9) | 48.6 (10.2)
  Depressive Problems | 58.5 (9.0) | 58.4 (8.3)

6. Secondary Outcome: Adolescent Quality of Life
Description: Pediatric Quality of Life (PedsQL) is a self-reported measure of diabetes-related quality of life in youth. Scaled scores range from 0-100, with higher scores indicating better quality of life.
Time Frame: 3 months
Population: Only adolescent participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 65
score on a scale | 67 (15) | 69 (14)

7. Secondary Outcome: Diabetes-related Family Conflict - Parent Report
Description: Diabetes-specific family conflict was measured with the Revised Diabetes Family Conflict Scale (DFCS), which consists of 19 items regarding how much adolescents and parents argue about diabetes management. Scores range from 19-57, with higher scores indicating higher levels of conflict.
Time Frame: 3 months
Population: Only maternal caregiver participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 69
score on a scale | 28.2 (4.9) | 28.8 (6.8)

8. Secondary Outcome: Diabetes-related Family Conflict - Adolescent Report
Description: Diabetes-specific family conflict will be measured with the Revised Diabetes Family Conflict Scale (DFCS), which consists of 19 items regarding how much adolescents and parents argue about diabetes management. Scores range from 19-57, with higher scores indicating higher levels of conflict.
Time Frame: 3 months
Population: Only adolescent participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 65
score on a scale | 30.1 (9.8) | 30.2 (10.7)

9. Secondary Outcome: Adolescent Diabetes Distress
Description: Problem Area in Diabetes - Teen (PAID-T) consists of 14 items measuring adolescents' diabetes distress. Scores range from 14-84, and scores of 44 or higher are considered clinically meaningful.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 65
score on a scale | 74 (30) | 64 (27)

10. Secondary Outcome: Diabetes Knowledge
Description: Revised Brief Diabetes Knowledge Test is a measure of parents' diabetes knowledge. It consists of 23 items that ask about diabetes-related information. Scores range from 0-23, with higher scores indicating greater diabetes knowledge.
Time Frame: 3 months
Population: Only maternal caregiver participants completed this measure.
Measure: Mean (Standard Deviation); unit: percentage of items correct
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 69
percentage of items correct | 69 (37) | 82 (27)

11. Secondary Outcome: Parental Involvement
Description: Collaborative Parent Involvement (CPI) is a 12-item scale completed by adolescents to assess parental involvement in diabetes care. Mean scores range from 1-5, with higher scores indicating more collaborative parental involvement.
Time Frame: 3 months
Population: Only adolescent participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 65
score on a scale | 4.1 (0.8) | 4.0 (0.9)

12. Secondary Outcome: Adolescent Adherence
Description: Self Care Inventory (SCI) is a 14-item measure completed by adolescents to assess their diabetes self-management behaviors. Mean scores range from 1-5, and higher scores indicate better adherence to the diabetes regimen.
Time Frame: 3 months
Population: Only adolescent participants completed this measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 60 | 65
score on a scale | 3.6 [2.9 to 4.0] | 3.7 [3.3 to 4.1]

13. Secondary Outcome: Quality of Parental Involvement
Description: Mothers and adolescents will participate in a videotaped conversation, which will be scored by objective raters using the Iowa Family Interaction Rating Scales (IFIRS). The collaborative parenting composite includes the following codes: Communication; Positive Reinforcement; and Child Centered. Scores on the collaborative parenting composite range from 3-27, with higher scores indicating higher levels of collaborative parenting. The overinvolved/intrusive parenting composite includes: Parental Influence; Intrusiveness; and Lecture/Moralize. Scores on the overinvolved scale range from 3-27, with higher scores indicating higher levels of observed behavior.
Time Frame: 6 months
Population: Analysis conducted if participants had baseline and 6 month videos.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication & Coping Intervention | Education & Check Ins
Number analyzed (Participants) | 27 | 27
score on a scale
  Collaborative Parent Behaviors | 14.8 (3.6) | 13.1 (3.6)
  Intrusive Parent Behaviors | 9.6 (4.2) | 9.9 (4.0)

ADVERSE EVENTS:
Time Frame: 1 year (study period)
Description: Only adolescent participants were assessed for adverse events. Participants' medical records were reviewed for any emergency department visits during the study project period (12 months). These were reviewed by the study endocrinologist to determine if they met the criteria for Diabetic Ketoacidosis (DKA).
  None of the adverse events were related to participation in the trial.
Arm/Group | Communication & Coping Intervention | Education & Check Ins
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 2/75 | 3/76
Other Adverse Events (participants affected / at risk) | 7/75 | 5/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Communication & Coping Intervention (N=75) | Education & Check Ins (N=76)
DKA (Endocrine disorders) | 2 (3) | 3 (8) — ED Visit for DKA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Communication & Coping Intervention (N=75) | Education & Check Ins (N=76)
Indicated Self-Harm or Suicidality (Psychiatric disorders) | 7 (9) | 5 (9) — Child endorsed the item "I deliberately try to hurt or kill myself" or "I think about killing myself" on the Youth Self Report measure. All events were followed up by the PI (a licensed clinical psychologist) and/or the clinic social worker.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT03818711/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT03818711/ICF_000.pdf